CLINICAL TRIAL: NCT01100216
Title: Human Laboratory Study of Smokeless Tobacco Products
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding expired prior to implementing subject recruitment.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2009NTLS097; 0911M74614 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Smokeless Tobacco
Keywords: smokeless tobacco; nicotine; snus; snuff; chewing tobacco; oral tobacco
MeSH Terms: conditions — Tobacco Use | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nicotine Lozenge (Active Comparator): 4 mg nicotine lozenge (LOZ
  Interventions: Other: Nicotine Lozenge
- Camel Snus Frost (Active Comparator)
  Interventions: Other: Camel Snus Frost
- Stonewall Spearment Tablet (Active Comparator)
  Interventions: Other: Stonewall Dissolvable Tobacco Pieces
- Skoal Wintergreen (Active Comparator)
  Interventions: Other: Skoal Wintergreen

INTERVENTIONS:
Other: Nicotine Lozenge — 4 mg for 12 days
  Other Names: Commit Nicotine Lozenge
  Arms: Nicotine Lozenge
Other: Stonewall Dissolvable Tobacco Pieces — 5.6 mg nicotine pieces for 12 days
  Other Names: Stonewall Spearmint Tablet
  Arms: Stonewall Spearment Tablet
Other: Camel Snus Frost — pouches, 6.2 mg nicotine, for 12 days
  Other Names: Camel Snus Frost Pouches
  Arms: Camel Snus Frost
Other: Skoal Wintergreen — Used at baseline (Days 1 and 2, 5-11) and then at every 7 day wash-out period.
  Other Names: Skoal
  Arms: Skoal Wintergreen

SUMMARY:
With the advent of restrictions on public smoking, the tobacco industry has introduced a variety of novel smokeless tobacco products (NSTP) to allow continued tobacco use. These products typically have lower tobacco-specific nitrosamines, carcinogens and nicotine than conventional smokeless products out on the market. No studies have compared the effects of NSTP and medicinal nicotine products (MNP) in smokeless tobacco users and whether some of the NSTP products may serve as a cessation tool for smokeless tobacco users. Our hypothesis is that the effects from these products will be directly related to their nicotine content and sensory effects. Products that produce greater effects on outcome measures may serve as potential cessation tools.

DETAILED DESCRIPTION:
Treatment will be a 3-period crossover study using Commit Nicotine Lozenge, Stonewall Disposable Tobacco Pieces and Camel Snus Frost Pouches. Each period will last 14 days with 11 days of product use and 1.5 days abstinence of all nicotine-containing products for a total of 10 weeks. Participants will begin the study by completing a baseline assessment on their own product, Skoal Wintergreen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be 20 male smokeless tobacco (SLT) users who are not seeking to quit (less than 5% of females use SLT.
* Subjects will be Skoal Wintergreen SLT users, since this is the most commonly used SLT that uses a mint-type flavorant.
* Subjects will have used SLT for at least 1 year..
* Subjects will be English speaking and reading.
* Provide written informed consent.

Exclusion Criteria:

* Subjects who have used other tobacco products (i.e., cigarettes, cigars) or nicotine products in past 6 months.
* Subjects who take medications that might affect the outcome of laboratory measures.
* Subjects with a history of major mood, thought, anxiety or attentional disorders.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Withdrawal Severity | Week 10
  Comparing withdrawal symptoms between the different products - 4 mg nicotine lozenge (LOZ), Camel Snus Frost (SNUS), Stonewall Spearmint Tablet (STAB), and Skoal Wintergreen (SKOL).

SECONDARY OUTCOMES:
Cognition Impairments | Week 10
  Comparing differences between the smokeless tobacco products - 4 mg nicotine lozenge (LOZ), Camel Snus Frost (SNUS), Stonewall Spearmint Tablet (STAB), and Skoal Wintergreen (SKOL).
Startle Response | Week 10
  Negative emotional responses to nicotine-relevant stimulant (based on physiologoical and electrophysiological measures, and self-reports of affective valence, arousal and control/dominance) differences between products - 4 mg nicotine lozenge (LOZ), Camel Snus Frost (SNUS), Stonewall Spearmint Tablet (STAB), and Skoal Wintergreen (SKOL).
Reinforcement | Week 10
  The break point (response workload at which subjects do not respond sufficiently to obtain a dosage of product in a defined time period) is expected to differ significantly between products - 4 mg nicotine lozenge (LOZ), Camel Snus Frost (SNUS), Stonewall Spearmint Tablet (STAB), and Skoal Wintergreen (SKOL).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Mooney, Ph.D., Principal Investigator — Dept. Psychiatry, University of Minnesota
Locations (1):
- Tobacco Research Center, Minneapolis, Minnesota, United States